CLINICAL TRIAL: NCT06457464
Title: Clinical Outcomes and Prognostic Factors in Patients With Multiple Myeloma in Assuit University Hospitals ( Prospective and Retrospective Study)
Brief Title: Clinical Outcomes and Prognostic Factors in Multiple Myeloma Patients
Status: Not yet recruiting | Type: Observational
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Amira Hassan Hassan Bakr, Doctor, Assiut University
Other Study IDs: COPFPMM
Record Dates: First submitted 2024-06-08; First posted 2024-06-13 (Actual); Last update posted 2024-06-13 (Actual); Status verified 2024-06

CONDITIONS: Multiple Myeloma
MeSH Terms: conditions — Multiple Myeloma | interventions — Drug Therapy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Drug: Chemotherapy — combination regimens including VCD (Velcade, cyclophosphamide, and dexamethasone ) or (MP) combination (melphalan and prednisolone) or VRD (Velcade, lenalidomide, dexamethasone) or VDT (Velcade, thalidomide, dexamethasone) or CRD (Cyclophosphamide, lenalidomide, dexamethasone ) or CDT (Cyclophosphamide, thalidomide, dexamethasone)

SUMMARY:
1. Description of the demographic, clinical, and laboratory characteristics of patients with MM admitted to the hematology unit of Assuit University Hospitals.
2. Determination of treatment outcomes and prognostic factors associated with survival rates.

DETAILED DESCRIPTION:
Multiple Myeloma MM (plasma cell myeloma) represents a malignant proliferation of plasma cells derived from B cells. Its median age of diagnosis is 52-61 years but is less common under 40 years. Males are affected more than females.

Diagnostic criteria for Multiple Myeloma:

1. Clonal bone marrow plasma cells or biopsy-proven bony or extramedullary plasmacytoma and any one of the following myeloma-defining events.
2. Evidence of one or more end-organ damage that can be attributed to the underlying plasma cell proliferative disorder specifically:

   * Hypercalcemia: serum calcium > 0.25mmol/l(>1 mg /dl) higher than the upper limit of normal or > 2.75mmol/l (>11mg/dl).
   * Renal insufficiency: creatinine clearance <40 ml per min or serum creatinine >177 µmol (>2 mg/dl) .
   * Anaemia : (hemoglobin value of < 10g/dl or hemoglobin > 2g/dl below the lower limit of normal
   * Bone lesions: one or more osteolytic lesions on skeletal radiography, CT or PET CT ∙ Any one or more of the following biomarkers of malignancy:

     * Clonal bone marrow plasma cells percentage > 60 %.
     * Involved: uninvolved serum-free light chain ratio ≥100.
     * >1 focal lesion on MRI studies. It causes many organ dysfunctions and symptoms such as renal failure, bony pains or fractures, anemia, susceptibility to infection, hypercalcemia, neurologic symptoms, and manifestation of hyperviscosity. It is characterized by the development of osteolytic lesions in the bone and involves the activation of osteoclasts with simultaneous suppression of new bone formation of osteoblast inhibition Bone pain is the most common symptom. Other presentations are anemia, hypercalcemia, renal failure, weight loss. Rare features are cord compression and CNS involvement.

The MM stage at presentation was documented according to the International Staging System (ISS) scoring and Durie-Salmon.

Over the last few decades, the management of MM has included chemotherapy: combination regimens including VCD (Velcade, cyclophosphamide, and dexamethasone ) or (MP) combination (melphalan and prednisolone) or VRD (Velcade, lenalidomide, dexamethasone) or VDT (Velcade, thalidomide, dexamethasone) or CRD (Cyclophosphamide, lenalidomide, dexamethasone ) or CDT (Cyclophosphamide, thalidomide, dexamethasone).

Then Follow-up will be for the patients after receiving their treatment for at least 18 months regarding response and survival analysis. and the novel therapies have significantly improved outcomes Autologous stem cell transplantation (ASCT) is an essential treatment strategy in the management of MM in young and fit patients.

In this study, we will present data of MM patients at the hematology unit in Assuit University hospitals from the year {2015:2025} including the demographic details, clinical presentations, laboratory features, treatment provided, response, and outcomes. We intended to explore the current situation of MM management, including the variety of drugs used and their responses, and patients undergoing ASCT and its outcome.

ELIGIBILITY:
Inclusion Criteria:

Patients ≥ 18 years old diagnostic as MM with Eastern Cooperative Oncology Group performance status(ECOG) Performance Status (0-2)

Exclusion Criteria:

Patients with poor performing status unfit to receive chemotherapy with ECOG PS > 2

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Sample size was calculated using Epi- Info7. According to results of previous study. Based on this percentage, confidence limits of 5% and a confidence level of 90%, the sample needed for the study was estimated to be about 97 patients.
Sampling Method: Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2024-07-01 (Estimated); Primary Completion 2025-08-01 (Estimated); Study Completion 2025-10-01 (Estimated)

PRIMARY OUTCOMES:
variety of drugs used and their responses, and pateints | baseline
  examine the current state of multiple myeloma management, including the variety of drugs used and their effectiveness, as well as the outcomes for patients undergoing autologous stem cell transplantation (ASCT).

REFERENCES:
- [Background] Kyle RA, Gertz MA, Witzig TE, Lust JA, Lacy MQ, Dispenzieri A, Fonseca R, Rajkumar SV, Offord JR, Larson DR, Plevak ME, Therneau TM, Greipp PR. Review of 1027 patients with newly diagnosed multiple myeloma. Mayo Clin Proc. 2003 Jan;78(1):21-33. doi: 10.4065/78.1.21. PMID 12528874
- [Background] Shin J, Koh Y, Youk J, Kim M, Kim BS, Choi CW, Sung HJ, Park Y, Yoon SS, Kim I. Clinicopathological characteristics of extremely young Korean multiple myeloma patients: therapeutic implications. Korean J Intern Med. 2017 Jul;32(4):722-730. doi: 10.3904/kjim.2016.256. Epub 2017 Jun 26. PMID 28651310
- [Background] Greipp PR, San Miguel J, Durie BG, Crowley JJ, Barlogie B, Blade J, Boccadoro M, Child JA, Avet-Loiseau H, Kyle RA, Lahuerta JJ, Ludwig H, Morgan G, Powles R, Shimizu K, Shustik C, Sonneveld P, Tosi P, Turesson I, Westin J. International staging system for multiple myeloma. J Clin Oncol. 2005 May 20;23(15):3412-20. doi: 10.1200/JCO.2005.04.242. Epub 2005 Apr 4. PMID 15809451
- [Background] Richardson PG, Hideshima T, Anderson KC. Bortezomib (PS-341): a novel, first-in-class proteasome inhibitor for the treatment of multiple myeloma and other cancers. Cancer Control. 2003 Sep-Oct;10(5):361-9. doi: 10.1177/107327480301000502. PMID 14581890